CLINICAL TRIAL: NCT05769699
Title: Serum Biomarkers in Parkinson's Disease at Different Stages
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 4687
Record Dates: First submitted 2023-02-28; First posted 2023-03-15 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-02

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Biomarkers (Experimental)
  Interventions: Procedure: blood sample

INTERVENTIONS:
Procedure: blood sample — blood sample

SUMMARY:
* Determine clinical characteristics of parkinsonian patients in various stages of disease;
* Measure peripheral neurodegeneration, synaptic, and inflammation biomarkers in a population of parkinsonian patients at various stages of disease.
* Measure vesicular neurodegeneration, synaptic and inflammation biomarkers

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with idiopathic PD according to Movement Disorders Society (MDS) criteria;
* Age: 18-80 years;
* Signature of informed consent to participate in this study

Exclusion criteria.

* Women pregnant
* Inflammatory or autoimmune diseases

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-02-10 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Determine clinical characteristics of parkinsonian patients in various stages of disease | 3 years
  Determine clinical characteristics of parkinsonian patients in various stages of disease by means of MDS-UPDRS score changes.
Determine clinical characteristics of parkinsonian patients in various stages of disease | 3 years
  Determine clinical characteristics of parkinsonian patients in various stages of disease by means of NMS score changes.
Determine biooogical characteristics of parkinsonian patients in various stages of disease | 3 years
  dosage of serum IL-1b, IL6, IL-5, IL-4, IL17, TNFa, IFNg, IL10, total-alpha-synuclein, NfL, BDNF (ng/ml for all)

CONTACTS AND LOCATIONS:
Locations (1):
- Flavia Torlizzi, Roma, Italy